CLINICAL TRIAL: NCT02251756
Title: Performance of Different Application Regimens of ACTINICA® on Protection From UVR-induced Erythema After One Day of Sun Exposure in Fair-skinned Healthy Subjects.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RD.03.CIP.29114; ID RCB: 2014-A00491-46 (Other: French Health Authority (ANSM))
Record Dates: First submitted 2014-09-25; First posted 2014-09-29 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2014-09

CONDITIONS: Healthy Subjects, Male or Female, of 18-60 Years Old, With Phototype I, II or III, Not Pre-treated/Pre-protected Skin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Actinica, 0.8 mg/cm2, 1application (Experimental): Actinica, 0.8 mg/cm2, 1application over one day of sun exposure
  Interventions: Device: Actinica, 0.8 mg/cm2, 1 application
- Actinica, 0.8 mg/cm2, 2 applications (Experimental): Actinica, 0.8 mg/cm2, 2 applications over one day of sun exposure
  Interventions: Device: Actinica, 0.8 mg/cm2, 2 applications
- Actinica, 2 mg/cm2, 1 application (Experimental): Actinica, 2 mg/cm2, 1 application over one day of sun exposure
  Interventions: Device: Actinica, 2 mg/cm2, 1 application
- Actinica, 2 mg/cm2, 2 applications (Experimental): Actinica, 2 mg/cm2, 1 application over one day of sun exposure
  Interventions: Device: Actinica, 2 mg/cm2, 2 applications

INTERVENTIONS:
Device: Actinica, 0.8 mg/cm2, 1 application
  Arms: Actinica, 0.8 mg/cm2, 1application
Device: Actinica, 0.8 mg/cm2, 2 applications
  Arms: Actinica, 0.8 mg/cm2, 2 applications
Device: Actinica, 2 mg/cm2, 1 application
  Arms: Actinica, 2 mg/cm2, 1 application
Device: Actinica, 2 mg/cm2, 2 applications
  Arms: Actinica, 2 mg/cm2, 2 applications

SUMMARY:
Study objective To assess the performance of different application regimens of Actinica® on protection from UV rays-induced erythema throughout 1 day of sun exposure in fair-skinned healthy subjects (phototype I to III).

Study centers A total of 20 subjects will be enrolled in 1 site in France.

Methodology This will be a monocentre, randomised, controlled, investigator-blind, intra-individual comparative clinical investigation.

There will be a total of 6 visits for each subject. Each subject will participate for a period of maximum 35 days.

Study population Healthy subjects, male or female, at least 18-60 years old, with phototype I, II or III, not pre-treated/pre-protected skin, meeting specific inclusion/exclusion criteria.

The clinical investigation will be conducted in 2 parts.

Part 1 - SPF determination:

To determine the SPF of Actinica® with application of two different amounts (0.8 and 2 mg/cm2).

Part 2 - Sun exposure:

To assess the performance of the different application regimens of Actinica® on protection from UVR-induced erythema throughout 1 day of sun exposure.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18-60 years of age,
2. Subject with Phototype I, II or III,
3. Subject with individual typology angle (ITA) 28-70°,
4. Subject with healthy skin / not tanned on the back,

Exclusion Criteria:

1. Subject with obvious skin cancer forms within the test areas, 2. Subject with hairs on the treated area that might interfere with clinical investigation assessments, 3. Subjects who have performed sun bathing at least four months before enrolment, 10. History of sun allergy / Mallorca acne, active photo induced or photo aggravated disease, or abnormal response to the sun (e.g., photosensitive dermatoses, polymorphic light eruption, solar urticaria, systemic lupus erythematosus, or dermatomyositis).

11. The subject has received, applied or taken the forbidden treatments within the specified time frame prior to the Day 0 visit (list available on request)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-07; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
erythema score | Part 2 -Day 1

CONTACTS AND LOCATIONS:
Locations (1):
- Nice, France